CLINICAL TRIAL: NCT06391255
Title: Reference Values for Gastric Emptying Scintigraphy After Bariatric Surgery
Acronym: SCATTER
Status: Enrolling by invitation | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-2345
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Gastric Emptying; Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal weight loss group: TWL between 25% and 35%
  Interventions: Other: scintigraphy

INTERVENTIONS:
Other: scintigraphy — oesophageal and gastric emptying

SUMMARY:
Oesophageal and gastric scintigraphy evaluates the function of the gastrointestinal system including variables such as oesophageal transit and gastric emptying (GE). Some variables are known to change after bariatric surgery. In patients that have symptoms of pain or nausea after bariatric surgery, oesophageal and gastric scintigraphy plays an important role in determining the nature of symptoms and is necessary for adequate treatment. However, literature on reference values in the bariatric population are scarce. At this moment, quantitative evaluation of the scintigraphy cannot be performed and conclusions are based on visual interpretation. There is a need for a standardised scintigraphy protocol for the population that underwent bariatric surgery taking into account the changed anatomy and physiology. Then, reference values that describe the oesophageal transit and GE assessed using scintigraphy have to be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years;
* RYGB or SG as primary bariatric surgery;
* A 2 year post-operative period without significant peri-operative or postoperative complications that could affect oesophageal transit, GE, or weight loss;
* "Normal" weight loss, according to our expectations (25% < TWL < 35%);
* Participants must be able to adhere to the study visit schedule and protocol requirements;
* Participants must be able to give informed consent (IC) prior to any study procedures;
* Willing to be informed about incidental findings of pathology and approving of reporting this to their general physician.

Exclusion Criteria:

* Pre-existent oesophageal or gastric motility disorders, dysphagia, reflux, dumping syndrome, (postprandial) abdominal pain, neurological or metabolic conditions that significantly affect oesophageal or gastric motility;
* When using proton pump inhibitors (PPI) or H2-antagonists, the inability to stop using them for 3 days;
* Using opioids;
* Previous oesophago-gastric surgery, other than bariatric surgery;
* Unable to stop smoking for 24h;
* Pregnancy or breast-feeding;
* Patients with a drug or alcohol addiction;
* Gluten intolerance;
* Intolerance to tracer ingredients;
* Participating in another scientific study at the same time, if this study interferes with the current study in any way.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, we will include 50 patients who underwent bariatric surgery (RYGB and SG), with uncomplicated procedure, postoperative period of two years and "normal" weight loss (25% < TWL < 35%). Participants are required to have an uncomplicated post-operative procedure and "normal" weight loss as GE might be connected to complications and/or weight loss results. Duration of inclusion period will be 2024-2025.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
reference values for RYGB and GS patients | 2-3 years
  gastric emptying (T1/2 [min], retention [%/min], caloric emptying [cal/min], GE curve over time)
to describe SPECT/CT images and determine its benefit for anatomical correlation in asymptomatic (reference) and symptomatic population. | 2-3 years
to define reference values for RYGB- and SG-patients for oesophageal scintigraphy after bariatric surgery using an optimised protocol; | 2-3 years
  transit time [min], emptying rate [%/min]

SECONDARY OUTCOMES:
to explore the correlation of GE and oesophageal transit, and weight loss results or symptoms, using prospective data from this study and retrospective data from symptomatic patients and similar studies previously | 2-3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands